CLINICAL TRIAL: NCT03389698
Title: Developing Advanced Blood-Brain Barrier Permeability Imaging for Early Alzheimer's Disease
Brief Title: Developing Advanced Blood-Brain Barrier Permeability Imaging for Early AD
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 17-01336
Record Dates: First submitted 2017-12-26; First posted 2018-01-03 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — gadobutrol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Cohort A: Cognitively normal control participants aged 20 - 40 years. Participants will undergo a 3T brain scan that will last up to 60 minutes using the GRASP DCE-MRI sequence performed during the first 21 minutes of scan time.
  Interventions: Device: GRASP Dynamic Contrast-Enhanced (DCE) MRI; Device: 3T Brain Scan; Drug: Gadolinium-based Contrast Agent (GBCA) for MRI
- Cohort B: Cognitively normal control participants aged 65 - 85 years. Participants will undergo a 3T brain scan that will last up to 60 minutes using the GRASP DCE-MRI sequence performed during the first 21 minutes of scan time.
  Interventions: Device: GRASP Dynamic Contrast-Enhanced (DCE) MRI; Device: 3T Brain Scan; Drug: Gadolinium-based Contrast Agent (GBCA) for MRI
- Cohort C: Amnestic mild cognitive impairment (aMCI) patients aged 65 and older. Participants in Cohort C will be matched by age and gender to participants in Cohort B. Participants in Cohort C will undergo a 3T brain scan that will last up to 60 minutes using the GRASP DCE-MRI sequence performed during the first 9 minutes of scan time.
  Interventions: Device: GRASP Dynamic Contrast-Enhanced (DCE) MRI; Device: 3T Brain Scan; Drug: Gadolinium-based Contrast Agent (GBCA) for MRI

INTERVENTIONS:
Device: GRASP Dynamic Contrast-Enhanced (DCE) MRI — Golden-angle Radial Sparse Parallel (GRASP) DCE MRI is an MRI sequence designed to improve spatial and temporal resolution while enabling retrospective reconstruction with flexible temporal resolution.
Device: 3T Brain Scan — Up to 60 minutes, a portion of which uses the GRASP DCE-MRI sequence.
Drug: Gadolinium-based Contrast Agent (GBCA) for MRI — Gadavist/Gadobutrol is a gadolinium-based contrast agent indicated for intravenous use in diagnostic magnetic resonance imaging (MRI) in adults and children (2 years of age and older) to detect and visualize areas with disrupted blood brain barrier (BBB) and/or abnormal vascularity of the central nervous system.
  Other Names: Gadavist/Gadobutrol

SUMMARY:
Aging is the primary risk factor in aging-related dementia. An important initiating factor for the development and progression of cognitive impairment is disruption of the blood-brain barrier (BBB). BBB plays an important role in maintaining normal brain homeostasis and protecting neural tissues from toxins. It is hypothesized that such changes known to be common in aging and can be an early process that precedes Alzheimer's Disease (AD). The microvascular changes related to subtle BBB disruption can be measured with permeability-surface area (PS) derived from GRASP DCE-MRI acquired less than 10 minutes, and the patterns of increased PS in normal and abnormal aging are different.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that have been diagnosed with aMCI ages 65-85

Exclusion Criteria:

* Pregnant, planning to get pregnant, or nursing.
* Claustrophobia
* Cardiac pacemaker
* Intracranial clips, metal implants, unremovable jewelries, metal in eyes.
* History or presence of any other major medical, neurologic or psychiatric conditions, such as Alzheimer's diseases, Parkinson's diseases, and stroke.
* Renal or liver disease as this may cause concerns related to Gad-based contrast agent
* Allergy to the contrast agent Gadolinium

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy cognitively normal control subjects of both age cohorts will be recruited by the study coordinator from (i) a pool of established volunteer subjects at NYU Langone Health who previously participated in research and who have agreed to be contacted about future research, (ii) Health Insurance Portability and Accountability Act of 1996 (HIPAA)-compliant databases such as RedCap and DataCore, and (iii) individuals who have contacted NYU to express interest in participating in research as a healthy volunteer.
  Subjects with aMCI will be recruited by Dr. Wisniewski from an ongoing NIH-funded large grant at NYU Barlow Center.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2023-07-11 (Actual)

PRIMARY OUTCOMES:
Permeability Surface Area (PS) as Measured by GRASP DCE-MRI Sequence | Up to 21 Minutes
  PS is measured by quantifying the contrast agent flow through blood vessel walls per unit volume of brain while accounting for the blood flow rate in the vessel.
Blood-Brain Barrier (BBB) Permeability as Measured by GRASP DCE-MRI Sequence | Up to 21 Minutes
  Golden-angle Radial Sparse Parallel (GRASP) dynamic contrast-enhanced (DCE) MRI sequence will be collected for the quantification of subtle BBB leakage throughout the brain.

CONTACTS AND LOCATIONS:
Overall Officials: Yulin Ge, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States